CLINICAL TRIAL: NCT03693898
Title: MR in Patients With Neuromuscular Diseases
Brief Title: MR in Patients With Collagen VI Related Myopathies
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruth Salim (Other)
Responsible Party: Sponsor-Investigator, Ruth Salim, Medical student, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: H-18023049
Record Dates: First submitted 2018-10-01; First posted 2018-10-03 (Actual); Last update posted 2018-10-10 (Actual); Status verified 2018-10

CONDITIONS: Bethlem Myopathy; Ullrich Disease
MeSH Terms: conditions — Bethlem myopathy; Scleroatonic muscular dystrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Persons with collagen VI defect (Other): Observational
  Interventions: Other: Observeational

INTERVENTIONS:
Other: Observeational — No intervention, observational

SUMMARY:
Collagen VI-related diseases include Bethlem myopathy and Ulrich dystrophy. They are both caused by decreased levels or a lack of collagen VI. The first symptoms can be present at birth as joint laxity and hypotonic muscles; often seen with luxation of the hip and scoliosis. During childhood, patients may develop contractures of fingers, wrists, elbows and ankles. Muscle weakness often appears in childhood to early adulthood and is progressive. It often results in walking difficulties.

There is no treatment available for Behtlem and Ulrich dystrophies.

The primary aim of this study is to investigate the pattern of involved muscles, the function and quality of the muscles and the disease severity using MRI.

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* confirmed Bethlem myopathy or Ulrich disease

Exclusion Criteria:

* All contraindications for undergoing an MRI scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2019-05-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Muscle fat fraction | One MRI scan pr subject (exam lasts approximately 60 min)
  The Dixon MRI will be used to quantify the fat fraction in skeletal muscle

SECONDARY OUTCOMES:
Muscle strength | Exam lasts approximately 40-60 min
  MRC in order to test specific muscles in the subjects

CONTACTS AND LOCATIONS:
Overall Officials: John Vissing, Prof., MD, Study Director — CNMC, Rigshospitalet
Locations (1):
- Copenhagen Neuromuscular Center, Copenhagen, Østerbro, Denmark